CLINICAL TRIAL: NCT00932659
Title: Characterization of Cardiac Arrhythmias in End Stage Kidney Disease Patients on Hemodialysis Using an Implantable Continuous Cardiac Rhythm Monitoring Device: A Pilot Study
Brief Title: Continuous Cardiac Arrhythmia Monitoring in Hemodialysis Patients
Acronym: CARE-ESRD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00012031
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-02

CONDITIONS: Arrhythmias, Cardiac
Keywords: End-Stage Renal Disease; Hemodialysis; Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients: This is a single arm observational study. The single arm consists of adult hemodialysis patients without a prior history of cardiac arrhythmias who will be implanted with a continuous cardiac monitoring device (REVEAL, Medtronic) for an FDA approved indication.
  Interventions: Device: continuous cardiac monitoring device (REVEAL, Medtronic)

INTERVENTIONS:
Device: continuous cardiac monitoring device (REVEAL, Medtronic) — hemodialysis patients without a prior history of cardiac arrhythmias will undergo implantation of a continuous cardiac monitoring device, and will undergo 6 months of follow-up

SUMMARY:
Hemodialysis patients have a rate of fatal arrhythmias that is 40 times greater than the general population, but the causes and types of fatal arrhythmias they experience is unclear. The purpose of this prospective observational cohort study is to capture and characterize occult arrhythmias which occur in hemodialysis patients over a 6 month period. After informed consent and baseline assessment, 30 adult hemodialysis patients without a prior history of cardiac arrhythmias will undergo implantation of a continuous cardiac monitoring device (REVEAL, Medtronic). Three followup visits will be scheduled to download device data and quantify the number of potentially malignant arrhythmias which occur in study subjects during the 6 month period. Additionally, captured events will be monitored remotely via regular patient initiated transmission of device data every 2 weeks. Any serious occult arrhythmias detected will be immediately acted upon with a predefined management algorithm. Descriptive data and simple proportions will be used to describe the incidence and types of arrhythmias among the study cohort. Risks of this study include 1) potential loss of patient confidentiality 2) risks related to insertion of device including pocket hematoma, device infection, pain and discomfort secondary to procedure. These will be minimized by strict security measures to protect each patient's protected health information (PHI), preprocedural screening and insertion of monitoring devices by highly trained operators, and frequent careful direct patient followup.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* ESRD receiving hemodialysis for at least 3 months

Exclusion Criteria:

* Inability to give informed consent
* Pre-existing implantable cardiac device (pacemaker or ICD) or imminent device implantation
* Imminent renal transplantation
* Life expectancy < 1yr
* PT-INR or aPTT > 1.7 upper limit of normal (ULN) or history of bleeding diathesis
* Unstable medical condition as deemed by primary nephrologist or study staff
* Known sustained ventricular tachycardia due to non-reversible cause.
* Active infection
* Known atrial fibrillation
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke hemodialysis patients with end stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sana Al-Khatib, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Huikuri HV, Castellanos A, Myerburg RJ. Sudden death due to cardiac arrhythmias. N Engl J Med. 2001 Nov 15;345(20):1473-82. doi: 10.1056/NEJMra000650. No abstract available. PMID 11794197
- [Background] Al-Khatib SM, Sanders GD, Bigger JT, Buxton AE, Califf RM, Carlson M, Curtis A, Curtis J, Fain E, Gersh BJ, Gold MR, Haghighi-Mood A, Hammill SC, Healey J, Hlatky M, Hohnloser S, Kim RJ, Lee K, Mark D, Mianulli M, Mitchell B, Prystowsky EN, Smith J, Steinhaus D, Zareba W; Expert panel participating in a Duke's Center for the Prevention of Sudden Cardiac Death conference. Preventing tomorrow's sudden cardiac death today: part I: Current data on risk stratification for sudden cardiac death. Am Heart J. 2007 Jun;153(6):941-50. doi: 10.1016/j.ahj.2007.03.003. PMID 17540194
- [Background] Goldenberg I, Moss AJ, McNitt S, Zareba W, Andrews ML, Hall WJ, Greenberg H, Case RB; Multicenter Automatic Defibrillator Implantation Trial-II Investigators. Relations among renal function, risk of sudden cardiac death, and benefit of the implanted cardiac defibrillator in patients with ischemic left ventricular dysfunction. Am J Cardiol. 2006 Aug 15;98(4):485-90. doi: 10.1016/j.amjcard.2006.03.025. Epub 2006 Jun 19. PMID 16893702
- [Background] Herzog CA. Cardiac arrest in dialysis patients: approaches to alter an abysmal outcome. Kidney Int Suppl. 2003 May;(84):S197-200. doi: 10.1046/j.1523-1755.63.s84.17.x. PMID 12694343
- [Background] Herzog CA. Can we prevent sudden cardiac death in dialysis patients? Clin J Am Soc Nephrol. 2007 May;2(3):410-2. doi: 10.2215/CJN.01130307. Epub 2007 Mar 27. No abstract available. PMID 17699443
- [Background] Lehrich RW, Pun PH, Tanenbaum ND, Smith SR, Middleton JP. Automated external defibrillators and survival from cardiac arrest in the outpatient hemodialysis clinic. J Am Soc Nephrol. 2007 Jan;18(1):312-20. doi: 10.1681/ASN.2006040392. Epub 2006 Dec 6. PMID 17151332
- [Background] USRDS Annual Data Report. Bethesda: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from June 2009 to August 2010
Groups:
- Single Arm: Hemodialysis Patients Implanted With REVEAL Device: adult hemodialysis patients without a prior history of cardiac arrhythmias
  continuous cardiac monitoring device (REVEAL, Medtronic) : hemodialysis patients without a prior history of cardiac arrhythmias will undergo implantation of a continuous cardiac monitoring device, and will undergo 6 months of follow-up
Period: Overall Study
Arm/Group | Single Arm: Hemodialysis Patients Implanted With REVEAL Device
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Hemodialysis Patients Implanted With REVEAL Device
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Significant Arrhythmia Detected
Time Frame: 6 months
Population: All patients enrolled were analyzed in this observational study.
Measure: Number; unit: participants
Arm/Group | Single Arm: Hemodialysis Patients Implanted With REVEAL Device
Number analyzed (Participants) | 8
participants | 0

2. Secondary Outcome: Number of Participants Experiencing a Peridialytic or Intradialytic Arrhythmias
Time Frame: 6 months
Population: all participants included
Measure: Number; unit: participants
Arm/Group | Single Arm: Hemodialysis Patients Implanted With REVEAL Device
Number analyzed (Participants) | 8
participants | 0

ADVERSE EVENTS:
Arm/Group | Single Arm: Hemodialysis Patients Implanted With REVEAL Device
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
This is the 1st study of an implantable cardiac monitor in HD patients. Despite minimally invasive device implantation,collaboration between cardiology and nephrology, a large population of available subjects, we were able to enroll only 8 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No